CLINICAL TRIAL: NCT04378257
Title: Efficacy of Therapist Guided e-Therapy Versus Self-Help Therapy on Psychological Distress Among Individuals in Oman During COVID-19 Pandemic: An Open-Label 12 - Weeks Randomized Controlled Trail
Brief Title: Efficacy of Therapist Guided e-Therapy Versus Self-Help Therapy on Psychological Distress Among Individuals in Oman During COVID-19 Pandemic
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sultan Qaboos University (Other)
Collaborators: The Research Council (Unknown); Oman Medical Specialty Board (Unknown)
Responsible Party: Principal Investigator, Mohammed Al Alawi, Principal Investigator, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/2020
Record Dates: First submitted 2020-05-02; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Depressive Symptoms; Generalized Anxiety
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist Guided E-Therapy (Experimental): The participants in this group will be allocated weekly sessions with a trained aboard certified clinical psychologist via a web-based e-therapy platform. The sessions will be conducted in the Arabic or English languages.
  Following sessions would focus on psychological first aid based on the following interventional tools:
  Cognitive Behavior Therapy (CBT)
  * Acknowledging emotions and normalizing current stress
  * Differentiate dysfunction versus distress (identify any debilitating thoughts/emotions if applicable)
  * Behavioral Activation Acceptance and Commitment Therapy (ACT)
  * Grounding, Breathing, Acceptance of emotions, and de-fusion
  Interventions: Behavioral: Therapist Guided E-Therapy
- Self-Help Therapy (Active Comparator): The participants in the control group will be supplied with an automatic weekly newsletter through E-mail containing self-help information and tips to cope with distress associated with COVID-19 in Oman. The information will mainly comprise of behavioral tips from principles of CBT and ACT focusing on positive cognitive reinforcement, strengthening relationships and mindfulness practice.
  Interventions: Behavioral: Self-Help Therapy

INTERVENTIONS:
Behavioral: Therapist Guided E-Therapy — The participants in this group will be allocated weekly sessions with a trained aboard certified clinical psychologist via a web-based e-therapy platform.The link will direct the participant directly to a screen where they will be able to see and interact with the psychologist once a week. The sessions will be conducted in the Arabic or English languages.Following sessions would focus on psychological first aid based on the following interventional tools:
  Cognitive Behavior Therapy (CBT)
  * Acknowledging emotions and normalizing current stress
  * Differentiate dysfunction versus distress (identify any debilitating thoughts/emotions if applicable)
  * Behavioral Activation Acceptance and Commitment Therapy (ACT)
  * Grounding, Breathing, Acceptance of emotions, and de-fusion
  Arms: Therapist Guided E-Therapy
Behavioral: Self-Help Therapy — The participants in the control group will be supplied with an automatic weekly newsletter through E-mail containing self-help information and tips to cope with distress associated with COVID-19 in Oman. The information will mainly comprise of behavioral tips from principles of CBT and ACT focusing on positive cognitive reinforcement, strengthening relationships and mindfulness practice. The participants will be requested to use this information to manage any distress that they might experience. On the sixth week, the participants in the control group will be assessed on their mood and anxiety symptoms. Participants will also be requested to provide information on other self-help remedies that participants used to improve or manage their functionality (example, access to other websites, communication with close friends or family etc.)
  Arms: Self-Help Therapy

SUMMARY:
Background:

COVID-19 (Corona Virus Disease 2019) is a virulent infectious disease with an incubation period ranging between 2-14 days. This highly contagious disease is caused by Sars-Cov-2 (Severe Acute Respiratory Syndrome Coronavirus 2). The number of people infected by COVID-19 has increased exponentially since January as a result of traveling and contact with COVID-19 infected individual. Initially, the seriousness of COVID-19 was not gauged properly until World Health Organization classified it as Pandemic type infectious disease and rapidly made plans actions to fight against it on 20 January, 2020. The uncertainty and low predictability of COVID-19 not only threaten people's physical health, but also affect people's mental health, especially in terms of emotions and cognition. As consequence of public emergency, with its economic health and social impacts, psychological repercussions among people are inevitable at the short and long term.

Importance and justify the study:

This study will assess the effectiveness of e therapy in treating anxiety and depression during a pandemic. This would be a novel way of providing therapy during crises

Hypothesis:

We hypothesize that compared to self-help email delivered therapy, the therapist guided e-Therapy is more efficacious in reducing the level of psychosocial stress among distressed individuals in Oman during COVID19.

Objective:

The aim of this study is to assess the efficacy of six weeks therapist guided e-Therapy versus Self-help e-mail delivered therapy on Psychological distress among random sample of individuals live in Oman during COVID 19 pandemic.

This study will recruit 60 participants from a list respondents to public survey who reported high levels of depression and anxiety, and randomize them to either therapist guided e-psychotherapy(intervention) or (control) self-help arms. Participants in the intervention arm will receive six sessions of therapist guided e therapy as described in the study schedule. Participants in the control arm will receive self-help psychotherapy contents similar to the intervention arm as detailed in the study schedule. Throughout the study, outcome and safety assessments will be conducted.

DETAILED DESCRIPTION:
COVID-19 (Corona Virus Disease 2019) is a virulent infectious disease with an incubation period ranging between 2-14 days. This highly contagious disease is caused by Sars-Cov-2 (Severe Acute Respiratory Syndrome Coronavirus 2). The number of people infected by COVID-19 has increased exponentially since January as a result of traveling and contact with COVID-19 infected individual. Initially, the seriousness of COVID-19 was not gauged properly until World Health Organization classified it as Pandemic type infectious disease and rapidly made plans actions to fight against this disease on 20 January, 2020. Ever since then, epidemic prevention was comprehensively upgraded and marked the real beginning of universal concern, indicating widespread impacts. The uncertainty and low predictability of COVID-19 not only threaten people's physical health, but also affect people's mental health, especially in terms of emotions and cognition. As consequence of public emergency, with its economic health and social impacts, psychological repercussions among people are inevitable at the short and long term. For instance, self-isolation and self-quarantine are often an unpleasant experiences for those who should endure them. Quarantine is the separation and restriction of movement of people who have potentially been exposed to a contagious disease to ascertain if they become unwell, so reducing the risk of them infecting other. This definition differs from isolation, which is the separation of people who have been diagnosed with a contagious disease from people who are not sick; however, the two terms are often used interchangeably, especially in communication with the public. Separation from loved ones, the loss of freedom, uncertainty over about the disease situation, financial consequences of not being at work, and boredom can have significant impact on the individuals. Furthermore, shortage of supply of basic needs, inadequate information/ misinformation and stigma of being infected are major concerns during these times. A number of studies studying stigma during times of pandemic showed the participants endorsed discrimination evident by others treating them differently: avoiding them, withdrawing social invitations, treating them with fear and suspicion, and making critical comments. In the literature, depression, anxiety and post-traumatic stress disorder are known sequalae of such pandemic in the past. Surge in suicide thoughts and hopelessness have been reported amid previous public health crisis.

With above being mentioned and given the paucity of literature from this part of the world, the researchers embark on studying the psychological impact of COVID-19 among Omani public and decipher the personal and socio-demographic characteristics shaping individual's resilience and psychological wellbeing. Those with high level of psychological distress will be invited to participate in 12 weeks randomized control trial of e-Therapy. Such endeavor would inform the public and policy maker to preemptively take the necessary steps in helping people during crisis to avoid major losses secondary to psychological degeneration.

Importance and justify the study:

This study will assess the effectiveness of e therapy in treating anxiety and depression during a pandemic. This would be a novel way of providing therapy during crises

Hypothesis:

We hypothesize that compared to self-help email delivered therapy, the therapist guided e-Therapy is more efficacious in reducing the level of psychosocial stress among distressed individuals in Oman during COVID19.

Objective:

The aim of this study is 1- To identify people with depression and anxiety symptoms during COVID-19 using GAD-7 AND PHQ-9 scales.

2- To assess the efficacy of six weeks therapist guided e-Therapy versus Self-help e-mail delivered therapy on Psychological distress among random sample of individuals live in Oman during COVID 19 pandemic.

Method Design and study site In this 12-week, open-label, comparative trial, participants will be randomized to receive either e-Therapy or self-help therapy, using a fixed randomization schedule allocating participant between the two treatment arms in a 1:1 ratio. This study will be conducted virtually using a secure encrypted video conference platform to deliver the e-Therapy to participants in intervention arm across Oman.

Allocation, concealment and randomization A software randomizer will be used to generate block randomization (block size is 6 ) in a 1:1 ratio to balance the number of the subjects in each arm . Block randomization is a commonly used technique in clinical trial design to reduce bias and achieve balance in the allocation of participants to treatment arms. Block randomization works by randomizing participants within blocks such that an equal number are assigned to each treatment. For example, given a block size of 4, there are 6 possible ways to equally assign participants to a block.

Participants allocation sequence either in intervention or control arm will be concealed from the study participants and the researchers before the beginning of the trial to avoid selection bias and it will be done through centralized service at the department of behavioural medicine. Each code will be given a sealed opaque envelope which will contain that participant's treatment allocation, and which will only be opened by research personnel not involved in the study or the process of data collection. All participants will have a code number allocated to them. As the design of this trial is open label, the participant and therapist who will conduct the therapy will be made aware of the intervention status after randomization finish. However, the outcome assessor,the person who will receive final outcome assessment e mails, will be blind to the participant's allocation.

Sample Size The sample size was calculated using nMaster 2.0. The Superiority hypothesis parallel clinical trial model was adopted to calculate the required sample size in each arm to achieve a mean effect size of Glass's Δ = 0.75, according to published literature of Therapist guided e-Therapy. Taking the power as 80% and 5% rate of type one error, the needed sample size will be 36 participants in each arm after considering 20% attrition rate.

Participants selection and eligibility Inclusion criteria

* All Omanis and Non-Omanis living in Oman, Male or female aging 18-65 years, with PHQ-9 or GAD -7 total scores ≥ 10
* Has access to the internet and video conferencing
* Able to participate in the trial and adhere to the trial protocol.
* Can provide a written informed consent to participate in the trial. Exclusion criteria
* Pre-existing mental disorders
* Diagnosis of moderate to severe intellectual disability.
* Presence of alcohol or other substance use disorders (except for nicotine or caffeine)
* Those who does not meet the inclusion criteria
* Those with suicidal or homicidal ideation at baseline. Intervention arm: Therapist Guided E-Therapy The participants in this group will be allocated weekly sessions with a trained aboard certified clinical psychologist via a web-based e-therapy platform. The psychologist will send an invitation e-link to the participant via e-mail prior to the scheduled meeting. The link will direct the participant directly to a screen where participants will be able to see and interact with the psychologist once a week. The sessions will be conducted in the Arabic or English languages.

The initial sessions would focus on building rapport and the focus would primarily be on the on-going events and experiences of the participants after the COVID-19 outbreak. Following sessions would focus on psychological first aid based on the following interventional tools:

Cognitive Behavior Therapy (CBT)

* Acknowledging emotions and normalizing current stress
* Differentiate dysfunction versus distress (identify any debilitating thoughts/emotions if applicable)
* Behavioral Activation Acceptance and Commitment Therapy (ACT)
* Grounding, Breathing, Acceptance of emotions, and de-fusion The final sessions would primarily focus on gathering data through the assessments and terminating the therapeutic relationship.

Control arm The participants in the control group will be supplied with an automatic weekly newsletter through E-mail containing self-help information and tips to cope with distress associated with COVID-19 in Oman. The information will mainly comprise of behavioral tips from principles of CBT and ACT focusing on positive cognitive reinforcement, strengthening relationships and mindfulness practice. The participants will be requested to use this information to manage any distress that they might experience. On the sixth week, the participants in the control group will be assessed on their mood and anxiety symptoms. Participants will also be requested to provide information on other self-help remedies that participants used to improve or manage their functionality (example, access to other websites, communication with close friends or family etc.)

Outcome Measures The Patient Healthcare Questionnaire (PHQ-9) is a self-administered measure used to make a tentative diagnosis of depression and monitor its severity. The PHQ-9 has been validated in a number of studies from different population ; ; . In Oman, Al-Ghafri et al examined the applicability of PHQ-9 among medical doctors. The cut-off score of 10 gave the best trade-off between a sensitivity of 80.6% and a specificity of 94.0%. In this study, cut off 10 was used to indicate the presence of significant depression S within the following classification.

The Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 consists of a self-report questionnaire that allows for the rapid detection of GAD . Participants are asked if they were bothered by anxiety related problems over the past two weeks by answering seven items on a 4-point scale. The total scores ranged from 0 to 21. At a cutoff score of 9, the GAD-7 had a sensitivity of 89 % and a specificity of 82 % for detecting GAD compared with a structured psychiatric interview. However, the validation of Arabic version of GAD-7 indicated that a cutoff score of 10 had the best trade-off between sensitivity and specificity. , Therefore, in the current study researchers take a total score of 10 and above as the cut-off for significant anxiety.

GAD-7 and PHQ-9 are available to healthcare providers completely free of charge. Pfizer Inc., the legal copyright holder, explicitly states that "no permission [is] required to reproduce, translate, display or distribute.

Data related to Age, gender, Martial status, Number of children, region in Oman, looking after elderly or sick person, highest qualification, , studying abroad, Doctor ( yes , no ), if yes specify what specialty , Nurse, Yes or No , if yes specify what area of practice, are you working in health care? Yes or No, if yes specify your type of work, employed ( Yes, No) if yes specify type of employment, financial strains yes or no , physical health problems yes or no , specify if yes, mental health problems yes or no , if yes specify, self-isolation Yes or No, self-quarantine Yes or No, coping strategies specify, e-mail address will be collected

Primary endpoint -Change in the mean scores of PHQ-9 and GAD-7 from baseline to the end of the study between the intervention and the control.

-Secondary endpoint - Proportion of subjects with Significant Psycho-Social distress (PHQ-9 total score ≥ 10 or GAD-7 total score ≥ 10) between the two arms

Recruitment, recruitment period and consent procedure The recruitment will be taking place over a period of 2 weeks from May 1st till May 14, 2020. Participants will be recruited randomly from list of online survey respondents with significant psychological distress in Oman. This survey was conducted by the current trial team during first two weeks of April 2020 and included 1539 respondents from different regions Oman. The prevalence of psychological distress among the trial sample was 30%. The research assistant will contact eligible participant by email and if they are interested and they will be briefed about the trial protocol. All interaction with the subjects including explanation and consenting will be carried out in private tele/video interview. Potential participant will receive a thorough explanation of the objectives, procedures and risks of this protocol of this trial that is appropriate to their level of understanding and comprehension .Based on the autonomy principal ,it is the full right of the subject to decline to participate or to withdraw from the study at any time without prejudice. After the consent form is explained to the participant and all questions have been answered, the participant can discuss their participation with the family members. After the consent is read and discussed with family, the participant will sign an electronic informed consent, the investigator with remind the patient that their contribution is fully voluntarily, and they can withdraw at any time.

Follow up visits and assessment procedures and Data management After baseline assessment and receiving 6 sessions of Therapist guided e-Therapy or Self-Help therapy, participant will be assessed for outcome measures at Week 6 and Week 12 by the sending then email link containing GAD-7 and PHQ-9. Otherwise, Over the first 6 weeks, each visit will include, checking the Consent, compliance with protocol and if any adverse effects. Data of each participant will receive a unique cod (serial number) .All data will be entered initially in to specified file for each subjects in every visit and then it will be transferred to Epi data sheet at the end of the visits.

ELIGIBILITY:
Inclusion Criteria:

* All Omanis and Non-Omanis living in Oman, Male or female aging 18-65 years, with PHQ-9 or GAD -7 total scores ≥ 10.
* Has access to the internet and video conferencing.
* Able to participate in the trial and adhere to the trial protocol.
* Can provide a written informed consent to participate in the trial.

Exclusion Criteria:

* Pre-existing mental disorders.
* Diagnosis of moderate to severe intellectual disability.
* Presence of alcohol or other substance use disorders (except for nicotine or caffeine).
* Those who does not meet the inclusion criteria.
* Those with suicidal or homicidal ideation at baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive symptoms measured by Patient Health Questionnaire-9 | 6-12 weeks
  Depressive symptoms will be measured with the Patient Health Questionnaire-9 (PHQ-9) instrument. The PHQ-9 is a nine item survey to assess depressive symptoms over the previous 2 weeks. The patient may answer "not at all" (scored as a 0) , "several days" (scored as a 1), "more than half the days" (scored as a 2), or "nearly every day" (scored as a 3) for each item. The range in total scores is from 0 (no depressive symptoms or best outcome) to 27 (severe depressive symptoms or worst outcome). The primary out come measure is to calculate the change in the mean scores of PHQ-9 from baseline to the end of the study between the intervention and the control.
Change in Anxiety symptoms measured by Generalized Anxiety Disorder-7 | 6-12 WEEKS
  The Generalized Anxiety Disorder 7-item scale is a 7- item self-report measure of generalized anxiety. Participants rate the frequency with which they experience anxiety-related symptoms on a scale of 0 (Not at all) to 3 (Nearly every day). Total scores range from 0-21 with higher scores indicating greater anxiety symptoms.
  The second primary out come measure is to calculate the change in the mean scores of GAD-7 from baseline to the end of the study between the intervention and the control.

SECONDARY OUTCOMES:
Proportion of subjects with Significant Depression | 6-12 weeks
  Proportion of subjects with Significant Depression (Defined as PHQ-9 total score ≥ 10 ) in each arm
Proportion of subjects with Significant Anxiety | 6-12 weeks
  Proportion of subjects with Significant Anxiety (Defined as GAD-7 total score ≥ 10 ) in each arm

REFERENCES:
- [Derived] Al-Alawi M, McCall RK, Sultan A, Al Balushi N, Al-Mahrouqi T, Al Ghailani A, Al Sabti H, Al-Maniri A, Panchatcharam SM, Al Sinawi H. Efficacy of a Six-Week-Long Therapist-Guided Online Therapy Versus Self-help Internet-Based Therapy for COVID-19-Induced Anxiety and Depression: Open-label, Pragmatic, Randomized Controlled Trial. JMIR Ment Health. 2021 Feb 12;8(2):e26683. doi: 10.2196/26683. PMID 33512323